CLINICAL TRIAL: NCT03324334
Title: Prevalence of Graves Disease in Patients With Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Khaleel, principal investigator, Assiut University
Other Study IDs: PGDUC
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with ulcerative colitis Interventions to be administered: Thyroid antibodies and Thyroid sonography
  Interventions: Diagnostic Test: Thyroid antibodies; Diagnostic Test: Thyroid sonography
- Control group: normal control subjects selected from general population at random Interventions to be administered: Thyroid antibodies and Thyroid sonography
  Interventions: Diagnostic Test: Thyroid antibodies; Diagnostic Test: Thyroid sonography

INTERVENTIONS:
Diagnostic Test: Thyroid antibodies — Thyroid antibodies: Antithyroperoxidase(Anti-TPO), Anti-thyroglobulin (anti-TG) to detect graves disease in study and control groups
Diagnostic Test: Thyroid sonography — Thyroid sonography to detect anatomical changes in thyroid

SUMMARY:
Graves disease in ulcerative colitis:

The connection between Graves disease and Inflammatory bowel disease is well known in the literature, but thyroid disorders have not been considered extra-intestinal manifestations of ulcerative colitis. In most cases, the diagnosis of thyroid disease has preceded that of Inflammatory bowel disease. Early studies have suggested a relationship between thyroid abnormalities and ulcerative colitis . But it is still uncertain whether the coexistence of Grave's and ulcerative colitis diseases is due to a specific reason or a coincidence.

DETAILED DESCRIPTION:
Graves disease in ulcerative colitis:

The connection between Graves disease and Inflammatory bowel disease is well known in the literature, but thyroid disorders have not been considered extra-intestinal manifestations of ulcerative colitis. In most cases, the diagnosis of thyroid disease has preceded that of Inflammatory bowel disease . Early studies have suggested a relationship between thyroid abnormalities and ulcerative colitis .But it is still uncertain whether the coexistence of Grave's and ulcerative colitis diseases is due to a specific reason or a coincidence.

Concomitant Graves disease and ulcerative colitis; In general, the pathophysiology of ulcerative colitis is associated with theTh2 cytokine phenotype, and there is increased Th2 activity in Graves disease .Therefore, both Graves disease and ulcerative colitis are associated with a Th1/Th2 imbalance, with a dominance of Th2 responses. reported on a 26-year-old female who had a flare-up of ulcerative colitis and hyperthyroidism that was successfully treated with infliximab. In addition, they reported that theTh1/Th2 imbalance was improved 2 weeks after the initiation of infliximab therapy. However, it is still unclear whether Graves disease is an extra intestinal manifestation of ulcerative colitis or not Restricted to ulcerative colitis only, we found OR significantly increased for Grave's disease.

Increasing evidence suggests that Grave's disease (GD), an autoimmune thyroid disease (AITD) that accounts for 60%-80% of hyperthyroidism cases, might be related to the abnormal genetic expressions, imbalance of immune responses, increased Th2 activity and overgrowth of intestinal bacteria. For instance, the prior literature showed that some genetic factors, such as Human leukocytic antigen , PTPN22 and CTLA4, were associated with Graves disease Other studies also observed that hyperthyroidism with autoimmune gastritis is usually accompanied with low acid production that may subsequently lead to an overgrowth of intestinal bacteria Therefore, it is plausible that hyperthyroidism might be one of the potential risk factors for ulcerative colitis, because both ulcerative colitis and hyperthyroidism are polygenic diseases and may share analogous mechanisms Furthermore, genetic pathways and Th2-dominant immunological responses could contribute to the association between ulcerative colitis and hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. seventy five patients who are diagnosed with ulcerative colitis who were admitted to Internal medicine department and who attend outpatient clinics in Assiut University Hospital will be involved in this study

Exclusion Criteria:

1. Patients with diabetes mellitus.
2. patients with a diagnosis of other than ulcerative colitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: seventy five patients who are diagnosed with ulcerative colitis who were admitted to Internal medicine department and who attend outpatient clinics in Assuit University Hospital will be involved in this study compared with 20 normal control subjects selected from general population at random
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with graves disease in ulcerative colitis | In 2 days
  By use of thyroid antibodies and thyroid sonography

CONTACTS AND LOCATIONS:
Overall Officials: Alaa K Hussein, MD, Principal Investigator — Assiut University,Faculty Of medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shizuma T. Concomitant Thyroid Disorders and Inflammatory Bowel Disease: A Literature Review. Biomed Res Int. 2016;2016:5187061. doi: 10.1155/2016/5187061. Epub 2016 Mar 3. PMID 27042663